CLINICAL TRIAL: NCT03921931
Title: Assessment of Retinal Photoreceptor Outer Segment Length With Optical Coherence Tomography Before and After Light Stimulation - a Pilot Study
Brief Title: Retinal Photoreceptor Outer Segment Length Before and After Light Stimulation - a Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Doreen Schmidl, Associate Professor, MD, PhD, Medical University of Vienna
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: OPHT-050418
Record Dates: First submitted 2019-04-04; First posted 2019-04-19 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-03

CONDITIONS: Macular Degeneration, Dry; Primary Open-angle Glaucoma
Keywords: light stimulation; retinal photoreceptors; light adaptation; functional optical coherence tomography; optophysiology; intrinsic optical signals
MeSH Terms: conditions — Geographic Atrophy; Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- healthy volunteers (Experimental): light stimulation
  Interventions: Other: White light stimulation
- primary open angle glaucoma patients (Experimental): light stimulation
  Interventions: Other: White light stimulation
- age-related macular degeneration patients (Experimental): light stimulation
  Interventions: Other: White light stimulation

INTERVENTIONS:
Other: White light stimulation — Stimulation of the retina with white light

SUMMARY:
It has been shown that reactions of human retinal photoreceptors to a light stimulus can be measured with custom-made, research prototype optical coherence tomography (OCT) systems. This can be used as a biomarker for the function of the photoreceptors. Due to the high technical demands on the system, however, the technique is currently not available for clinical purposes. In this pilot study a protocol to measure changes in retinal photoreceptor layer thickness before and after light stimulation shall be developed based on a commercial OCT system and newly developed algorithms. Other variables, such as circadian processes shall be investigated as well. After measurements in healthy volunteers, the protocol is planned to be applied in patients with primary open angle glaucoma (POAG) and age-related macular degeneration (AMD) to test for feasibility of the method in these patient groups.

ELIGIBILITY:
Inclusion Criteria:

* men and women aged over 18 years
* signed informed consent form
* ametropia below 3 diopters
* ability and willingness to follow instructions

for healthy volunteers:

* normal ophthalmologic findings

for primary open angle glaucoma patients (POAG):

* diagnosed POAG
* MD <= 10 dB

for age-related macular degeneration (AMD):

* diagnosed dry AMD
* diagnosed stage II or stage III AMD

Exclusion Criteria:

* Presence of any abnormalities preventing reliable measurements
* Ocular inflammation and ocular disease interfering with the study aims
* Use of photosensitizing medication (phototoxic drugs, photoallergic drugs) in the 3 months preceding the study
* Presence of any condition with the possibility of causing photosensitivity, including systemic lupus erythematosus SLE, Porphyria, Vitiligo, Xeroderma Pigmentosum and Albinism
* Presence of any form of epilepsy
* Ocular surgery in the 3 months preceding the study
* Pregnancy, planned pregnancy or lactating
* Any medical or surgical history, disorder or disease such as acute or chronic severe organic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2018-11-26 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Light stimulation | 1 day
  Optical path length changes between inner segment outer segment junction and retinal pigment epithelium (RPE) will be measured with OCT in 15 healthy volunteers, 10 POAG patients and 10 AMD patients before and after light stimulation

SECONDARY OUTCOMES:
Light stimulation of contralateral eye | 1 day
  Optical path length changes between inner segment outer segment junction and retinal pigment epithelium (RPE) will be measured with OCT in 15 healthy volunteers, 10 POAG patients and 10 AMD patients before and after light stimulation in the contralateral eye
Difference in photoreceptor layer thickness over the course of 8 hours | 8 hours
  Influence of circadian rhythm on the length of retinal photoreceptor outer segments
En face maps | 1 day
  test an algorithm for production of en face maps of retinal photoreceptor outer segment length

CONTACTS AND LOCATIONS:
Overall Officials: Doreen Schmidl, MD,PhD, Principal Investigator — Department of Clinical Pharmacology, Medical University of Vienna
Locations (1):
- Medical University of Vienna, Department of Clinical Pharmacology, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No